CLINICAL TRIAL: NCT06897501
Title: Incidence of Postoperative Vocal Cord Palsy Between Double-lumen Endobronchial Tube and Bronchial Blocker for Robot-assisted Esophagectomy: a Multicenter Randomized Controlled Trial
Brief Title: Postoperative Vocal Cord Palsy Between Double-lumen Endobronchial Tube and Bronchial Blocker for Robot-assisted Esophagectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Joo Ahn, Professor, Anesthesiologist, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SMC 2024-12-120
Record Dates: First submitted 2025-03-25; First posted 2025-03-27 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: One Lung Ventillation (OLV)
Keywords: robot-assisted esophagectomy; double-lumen endobronchial tube; bronchial blocker; vocal cord palsy
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- double-lumen endobronchial tube group (Active Comparator)
  Interventions: Device: double-lumen endobronchial tube
- bronchial blocker group (Experimental)
  Interventions: Device: bronchial blocker

INTERVENTIONS:
Device: bronchial blocker — Lung isolation for robot-assisted esophagectomy will be performed using bronchial blocker in this group.
  Arms: bronchial blocker group
Device: double-lumen endobronchial tube — Lung isolation for robot-assisted esophagectomy will be performed using double-lumen endobronchial tube in this group.
  Arms: double-lumen endobronchial tube group

SUMMARY:
The goal of this clinical trial is to investigate whether the use of bronchial blocker could reduce the incidence of postoperative vocal cord palsy than the use of double-lumen endobronchial tube in robot-assisted esophagectomy.

DETAILED DESCRIPTION:
Esophagectomy is a challenging surgery that usually requires one lung ventilation, and double-lumen endobronchial tubes and bronchial blockers are commonly used for one lung ventilation.

Successful resection of recurrent laryngeal nerve lymph nodes during esophagectomy is important to survival and prevention of cancer recurrence, but there is a risk of postoperative vocal cord palsy due to the recurrent laryngeal nerve injury during the resection.

Compared to a double-lumen endobronchial tube, the use of a bronchial blocker is expected to reduce the incidence of recurrent laryngeal nerve injury; however, few clinical studies compare the two devices in terms of the incidence of postoperative vocal cord palsy in robot-assisted esophagectomy.

Therefore, the researchers aimed to investigate whether the use of bronchial blocker could reduce the incidence of postoperative vocal cord palsy than the use of double-lumen endobronchial tube in robot-assisted esophagectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 or older
* American Society of Anesthesiologists physical status I - III
* Elective robot-assisted esophagectomy
* Any clinical stage of esophageal cancer
* Patients who need recurrent laryngeal nerve lymph nodes resection

Exclusion Criteria:

* Patients who diagnosed vocal cord palsy or damage before surgery
* Patients who need specific airway device due to airway problem
* History of thoracic surgery
* Emergency surgery
* Combined surgery with other department
* Pregnant or nursing women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative vocal cord palsy | On postoperative day 7 after robot-assisted esophagectomy
  On postoperative day 7, ENT doctor will performed the laryngoscopy exam to check the presence of vocal cord palsy.

SECONDARY OUTCOMES:
Number of resected recurrent laryngeal nerve lymph nodes | At the end of surgery
  Number of successfully resected recurrent laryngeal nerve lymph nodes will be counted at the end of surgery
Quality of one lung ventilation | during one lung ventilation
  during one lung ventilation, anesthesiologists will evaluate the degree (excellent, fair, poor) of lung collapse.
Surgical difficulty reported by surgeon | At the end of surgery
  Surgeon will report the surgical difficulty (easy, moderate, difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Ahn, MD PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chao YK, Li Z, Jiang H, Wen YW, Chiu CH, Li B, Shang X, Fang TJ, Yang Y, Yue J, Zhang X, Zhang C, Liu YH. Multicentre randomized clinical trial on robot-assisted versus video-assisted thoracoscopic oesophagectomy (REVATE trial). Br J Surg. 2024 Jul 2;111(7):znae143. doi: 10.1093/bjs/znae143. PMID 38960881
- [Background] Li B, Yang Y, Toker A, Yu B, Kang CH, Abbas G, Soukiasian HJ, Li H, Daiko H, Jiang H, Fu J, Yi J, Kernstine K, Migliore M, Bouvet M, Ricciardi S, Chao YK, Kim YH, Wang Y, Yu Z, Abbas AE, Sarkaria IS, Li Z; Cooperative Group of International Expert Consensus on Robot-assisted Esophagectomy for Esophageal Cancer. International consensus statement on robot-assisted minimally invasive esophagectomy (RAMIE). J Thorac Dis. 2020 Dec;12(12):7387-7401. doi: 10.21037/jtd-20-1945. No abstract available. PMID 33447428
- [Background] Palaczynski P, Misiolek H, Szarpak L, Smereka J, Pruc M, Rydel M, Czyzewski D, Bialka S. Systematic Review and Meta-Analysis of Efficiency and Safety of Double-Lumen Tube and Bronchial Blocker for One-Lung Ventilation. J Clin Med. 2023 Feb 27;12(5):1877. doi: 10.3390/jcm12051877. PMID 36902663